CLINICAL TRIAL: NCT00800709
Title: Changes of Biological Markers and Brain PET Imaging and Clinical Effects of Memantine for Patients With Moderate to Severe Alzheimer's Disease: a 24 Week Double-blind, Randomized, Placebo-Controlled Study
Brief Title: Memantine and Changes of Biological Markers and Brain PET Imaging in Alzheimer's Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shanghai Mental Health Center (Other)
Collaborators: H. Lundbeck A/S (Industry)
Responsible Party: Department of Psychogeriatrics, Shanghai Mental Health Center, Shanghai Mental Heath Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IIT_12484A
Record Dates: First submitted 2008-10-23; First posted 2008-12-02 (Estimated); Last update posted 2010-12-03 (Estimated); Status verified 2010-12

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer's Disease; tau protein; PET; Memantine
MeSH Terms: conditions — Alzheimer Disease; Frontotemporal Dementia | interventions — Memantine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Memantine (Experimental)
  Interventions: Drug: Memantine

INTERVENTIONS:
Drug: Memantine — Initially memantine 5mg/day, titrated within the first month to a maintenance dose of 20mg/day
  Other Names: Memantine hydrochloride

SUMMARY:
In AD, tau protein is abnormally hyperphosphorylated. Significant changes of hyperphosphorylated tau levels in CSF are found in AD patients. It has been shown in vitro that memantine can reverse abnormal hyperphosphorylation of tau in hippocampal neurons of rats. A statistically significant reduction of CSF phosphorylated tau at a preliminary 1-year follow-up was observed, from median 126 (interquartile range 107-153) to 108 (88-133) ng/l (p = 0.018). No statistically significant differences of total tau or Aβ42 were found (Gunnarsson MD, 2007).

FDG-PET has the unique ability to estimate the local cerebral metabolic rate of glucose consumption, thus providing information on the distribution of neuronal death and synapse dysfunction in AD in vivo (Herholz K. 2003). Synaptic dysfunction and loss induce a reduction in neuronal energy demand that results in decreased glucose metabolism. Hypometabolism in AD is thought to reflect loss of synaptic activity and density (Herholz K. 2003; Mielke R, et al. 1998).

Another biological markers such as inflammatory factor and APOEε4 also play a part in the onset of AD (Glodzik-Sobanska L, 2007).

DETAILED DESCRIPTION:
1. To investigate the effects of daily dosing of memantine for 24 weeks versus placebo on biological markers of subjects with Alzheimer's disease.
2. To investigate the effects of daily dosing of memantine for 24 weeks versus placebo on 18[F]-FDG-PET of brain in subjects with Alzheimer's disease.
3. To investigate the effects of daily dosing of memantine for 24 weeks versus placebo on cognitive function in subjects with Alzheimer's disease.
4. To investigate the effects of daily dosing of memantine for 24 weeks versus placebo on measures of behavior and activities of daily living of subjects with Alzheimer's disease.
5. To investigate the effects of daily dosing of memantine for 24 weeks versus placebo on short term memory.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent
2. Clinical diagnosis of Alzheimer's disease which meet the DSM-IV criteria.
3. Subject has moderate to severe Alzheimer's disease as defined by a MMSE score 4 to 20 inclusive at screening.
4. Hachinski Ischemia Score < 4 at screening.
5. Age ≥50 and ≤90 years.
6. Availability of a responsible and steady caregiver to ensure treatment compliance and provide information for assessments.

Exclusion Criteria:

1. Severe renal impairment.
2. History of seizures
3. Systolic blood pressure >160 or < 90 mmHg or diastolic blood pressure > 95 or < 60 mmHg at the time of screening.
4. Diagnosis of any concomitant life threatening illness.

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2008-07; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
biological markers of CSF | 24 weeks
18[F]-FDG-PET of brain | 24 weeks
cognitive function | 24 weeks

SECONDARY OUTCOMES:
behavior and activities of daily living | 24 weeks
short term memory | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Shifu Xiao, MD. PhD., Principal Investigator — Department of Psychogeriatrics，Shanghai Mental Health Center
Locations (1):
- Department of Psychogeriatrics，Shanghai Mental Health Center, Shanghai, Shanghai Municipality, China